CLINICAL TRIAL: NCT01180738
Title: Comparison of Short Bursts of Body Weight Supported Treadmill Training vs. Overground Walking Training in Persons With Chronic Stroke
Brief Title: Body Weight Supported Treadmill Training vs. Overground Walking Training in Persons With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephanie Miller (Other)
Collaborators: University of Indianapolis (Other); Richard L. Roudebush VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Stephanie Miller, Professor, University of Indianapolis
Organization: University of Indianapolis (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BWSTTvsOWT_UIndy
Record Dates: First submitted 2010-08-09; First posted 2010-08-12 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Difficulty Walking
Keywords: chronic stroke; walking training; rehabilitation; body weight supported treadmill training; physical therapy; balance
MeSH Terms: conditions — Stroke; Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Body weight supported treadmill training (Active Comparator)
  Interventions: Behavioral: Body weight supported treadmill training
- Overground walking training (Active Comparator)
  Interventions: Behavioral: Overground walking training

INTERVENTIONS:
Behavioral: Body weight supported treadmill training — Training will include 10 sessions over a 2 week period, each session with 30 minutes of walking on a treadmill using a body weight support system.
  Arms: Body weight supported treadmill training
Behavioral: Overground walking training — Training will include 10 sessions over a 2 week period, each session with 30 minutes of walking overground.
  Arms: Overground walking training

SUMMARY:
The purpose of this study is to compare two different walking training programs for persons with chronic stroke.

DETAILED DESCRIPTION:
Body weight supported treadmill training (BWSTT) and overground walking training (OWT) are two interventions commonly applied for enhancing gait and balance in patients with chronic stroke. BWSTT and OWT are often used by clinicians separately or in tandem. While various aspects of the two interventions have been investigated in the past, limited research has been conducted to compare the effects of the two interventions in patients with chronic stroke.

Longer training durations may not always be feasible due to limited reimbursement options, lack of clinic accessibility, or transportation restrictions for patients with chronic deficits following stroke. A short burst of training consisting of a ''booster''-like protocol may provide a convenient option for some patients with chronic stroke to improve necessary functional skills in a short period of time.

The primary purpose of this pilot study is to compare walking speed immediately and 3-months after a short-burst of body-weight support treadmill training (BWSTT) or overground walking training (OWT) for adults with chronic stroke. Twenty participants with chronic stroke will be recruited and screened to determine eligibility for the study. Participants will be randomly assigned to either BWSTT or OWT for 30 minutes, 5 days per week for 2 weeks. Outcome measures will include assessments of gait speed, endurance, walking pattern, fear of falling, balance confidence, anxiety, and activity and participation in daily life. Outcomes will be tested prior to (pre-test) and immediately after (post-test) the assigned intervention and again 3-months after completing the intervention (retention).

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 6 months post-stroke
* Single episode of stroke
* Between the ages of 21-80
* Able to walk with or without the use of an assistive device or orthoses
* Able to ambulate at a self-selected gait speed < 0.8 m/s as determined by the 10-meter comfortable walk test
* Medically stable with a physician release stating approval to enter an exercise program
* Able to follow at least two-step verbal instructions
* Available for the entire period of the study
* Able to travel to and from research measurement and intervention sessions

Exclusion Criteria:

* Currently receiving physical therapy services
* Co-morbidities or pre-existing cardiovascular conditions that would prohibit gait training and exercise
* Pre-existing neurological or current musculoskeletal conditions that would limit gait ability separate from the effects of stroke
* Complications from other health conditions that could influence walking
* Currently known to be pregnant

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Gait speed: measured with the comfortable 10-meter walk test | The outcome measure will be assessed at pre-test (within 1-week before beginning the intervention), post-test (within 1-week after completing the 2-week intervention period) and at retention (3-months following completion of the intervention).

SECONDARY OUTCOMES:
Gait endurance: measured with the 6-minute walk test; Fear of falling: measured with the Fear of Falling questionnaire and Falls Efficacy Scale-International | The outcome measures will be assessed at pre-test (within 1-week before beginning the intervention), post-test (within 1-week after completing the 2-week intervention period) and at retention (3-months following completion of the intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Combs, PT, PhD, NCS, Principal Investigator — University of Indianapolis, Krannert School of Physical Therapy, Indianapolis, IN; Arlene A Schmid, OTR, PhD, Principal Investigator — Co-Investigator, Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- University of Indianapolis, Krannert School of Physical Therapy, Indianapolis, Indiana, United States